CLINICAL TRIAL: NCT05018299
Title: A Randomized, Placebo Controlled, Double Blind Phase IIa Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Clinical Activity of Multiple Intravenous Doses of FB704A in Adults With Severe Asthma
Brief Title: Evaluate the Efficacy and Safety of FB704A in Adult With Severe Asthma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Oneness Biotech Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: FB704ACLIS-02
Record Dates: First submitted 2021-08-15; First posted 2021-08-24 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Severe Asthma
Keywords: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- FB704A placebo (Placebo Comparator): placebo
  Interventions: Biological: FB704A placebo
- FB704A (Experimental): Anti-IL6 antibody
  Interventions: Biological: FB704A

INTERVENTIONS:
Biological: FB704A placebo — Placebo
  Arms: FB704A placebo
Biological: FB704A — Anti-IL-6 antibody
  Arms: FB704A

SUMMARY:
This is a randomized, placebo controlled and double blind study to evaluate the safety, tolerability, pharmacokinetics, and clinical activity of FB704A in adult patients with severe asthma. The study comprised a 4-week screening period, a 8-week treatment period and a 12-week follow-up period.

DETAILED DESCRIPTION:
Approximately 20 subjects who meet the criteria for study entry are planned to be enrolled to the study. Eligible subjects will be randomized to receive placebo or FB704A in a 1:1 ratio, with an estimated 10 subjects per treatment arm.

Eligibility will be checked in patients with severe asthma during the 4-week screening period. Potential candidates should provide signed informed consent forms before starting the screening activities. The subjects will receive four dose of 4 mg/kg FB704A or placebo. The study drug will be administered as a 1-hour IV infusion.

Patients may administer Short-acting beta agonists (SABAs), such as albuterol as rescue medications as needed throughout the study.

Subjects will have site visits after receiving study drug for efficacy, safety, PK, and biomarker evaluation (see Study Flow Chart). Subjects who prematurely withdraw from the study will have an end of study (EOS) visit within 7 days.

Relative change in pre-bronchodilator FEV 1 , post-bronchodilator FEV 1, exhaled NO and asthma symptom s will be evaluated during the study.

ELIGIBILITY:
Inclusion Criteria:

1.18 to ≦75 years of age, either sex, any race. 2.Diagnosed as severe asthma based on 2020 GINA guideline. 3.An ACT score is <20. 4.Induced sputum neutrophil count ≧50% of total sputum cells during Screening. 5.Documented diagnosis of severe asthma within past 5 years. Additionally, subjects must have at least one of the following: a) ≧12% and/or 200 mL improvement in Forced Expiratory Volume in 1 second (FEV1) post-bronchodilator, OR b) airway hyperresponsiveness (e.g., positive methacholine challenge <8 mg/mL), OR c) within the past 24 months, airway variability with a ≧12% and 200 mL change in FEV1 between clinic visits outside of respiratory infections, documented prior to Visit 1, OR d) within the past 24 months, average daily PEF variability > 10% over a 2-week period, documented prior to Visit 1.

6.Nonsmoker or previous smoker with cumulative smoking history less than 10 pack-years (pack-year = 20 cigarettes smoked daily for 1 year). Previous smokers may not have smoked within 1 year prior to Screening. A smoker is defined as a subject who has taken inhaled nicotine containing products (e.g. cigarette, cigar, pipe), including e-cigarettes prior to screening.

7.Must not have had a severe asthma exacerbation of asthma for 4 weeks prior to Screening and must be on a stable medication regimen for asthma at least 4 weeks prior to Screening.

A Severe asthma exacerbation is defined as a deterioration of asthma leading to treatment for 3 days or more with systemic glucocorticoids or hospitalization or an emergency department visit leading to treatment with systemic glucocorticoids.

8.Must be willing to give written informed consent to participate in the study. 9.Must be capable of complying with the dosing regimen, adhere to the visit schedule, and participate in all treatment procedures, including sputum induction.

10.Female subject of childbearing potential must have a negative serum pregnancy test at Screening and must be using a medically acceptable, highly effective, adequate form of birth control (ie, failure rate <1% per year when used consistently and correctly) prior to Screening and agree to continue using it while in the study (Screening and Treatment Periods). Medically acceptable, highly effective forms of birth control are hormonal implants, oral contraceptives, medically acceptable prescribed intrauterine devices (IUDs), and monogamous relationship with a male partner who has had a vasectomy. Female subject who is not of childbearing potential must have a medical record of being surgically sterile (eg, hysterectomy, tubal ligation), or be at least 1 year postmenopausal. Absence of menses for at least 1 year will indicate that a female is postmenopausal. A female subject should be encouraged to continue using a highly effective method of birth control for 30 days following the end of treatment.

Male subject must agree to use an adequate form of contraception for the duration of the study and agree to have sexual relations only with women who use a highly effective birth control method.

Exclusion Criteria:

1.Chronic Obstructive Pulmonary Disease (COPD)/other relevant lung disease (other than asthma) 2.4 weeks prior to/or Screening: upper/lower respiratory tract infection 3.Screening: Inadequate amount or difficulty producing sputum 4.Screening: Sputum neutrophil count over 10 million/mL 5.Screening: peripheral blood neutrophil (PBN) count <2000/µL 6.Clinically significant chronic infectious disease(s) (eg, Human Immunodeficiency Virus [HIV], hepatitis B or C) 7.Allergy/sensitivity to study drug/excipients 8.Breast-feeding, pregnant/intends to become pregnant during study 9.Requiring mechanical ventilation for respiratory event within 6 months of Screening 10.Medical condition(s) (eg, hematologic, cardiovascular, renal, hepatic, neurologic, or metabolic) or medication that may interfere with effect of study medication 11.Within 30 days of Screening: any other investigational drug 12.Known history of active tuberculosis (TB) or evidence of tuberculosis infection as defined by a positive purified protein derivative (PPD) skin test and/or interferon-gamma release assay. The interferon-gamma release assay should be repeated in case of an indeterminate result 13.Active infection, including opportunistic infections, requiring systemic therapy within the past 2 weeks 14.A deep space infection within the past 2 years (including, but not limited to meningitis, epiglottitis, endocarditis, septic arthritis, fasciitis, abdominal or pleural abscess, or osteomyelitis) 15.History of diverticulitis, diverticulosis requiring antibiotic treatment, or other symptomatic lower gastrointestinal (GI) conditions that might predispose to perforations 16.Immunization with a live/attenuated vaccine within 4 weeks prior to treatment 17.Evidence of active malignant disease, malignancies diagnosed within the previous 5 years (including hematological malignancies and solid tumors, except basal and squamous cell carcinoma of the skin or carcinoma in situ of the cervix uteri that has been excised and cured) 18.Liver enzymes: alanine aminotransferase (ALT) and aspartate aminotransferase (AST) > 3x upper limit of normal 19.Serum bilirubin > 2x upper limit of normal 20.Low platelet count (<100,000/mm3) 21.Dyslipidemia. 22.Participation in any other clinical study. 23.Part of the staff personnel involved with the study. 24.Family member of investigational study staff.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2026-02-13 (Estimated); Study Completion 2026-05-08 (Estimated)

PRIMARY OUTCOMES:
Proportion of the number of Adverse Event reported during the treatment period | Day 57
  AE

SECONDARY OUTCOMES:
Change from baseline in blood neutrophil counts | Day 36, 57, 85, 113, and 141
  neutrophil counts
Change from baseline in sputum neutrophil counts | Day 57
  neutrophil counts
ACT score | Day 36, 57, 85, and 141
  The ACT Score > 19 means well controlled.
Change from baseline in Asthma control test (ACT) | Day 36, 57, 85, and 141
  The ACT Score > 19 means well controlled.
Percentage of patients achieving decrease in score by greater than or equal to 0.5 points on the ACQ 5 (with a minimal importance difference improvement) | week 4, 8, 12, and 20
  The Asthma symptom score and 5 item Asthma Control Questionnaire (ACQ 5) will be applied to evaluate the condition of asthma control. Subjects will perform the test.
Change from baseline in ACQ-5 | Day 36, 57, 85, and 141
  The Asthma symptom score and 5 item Asthma Control Questionnaire (ACQ 5) will be applied to evaluate the condition of asthma control. Subjects will perform the test.
Change from baseline in AQLQ | Day 36, 57, 85, and 141
  Standardized Asthma Quality of Life Questionnaire (AQLQ) will be applied to evaluate the asthma specific quality of life.
Change from baseline in pre-bronchodilator FEV1 , post-bronchodilator FEV1, exhaled NO and asthma symptoms | Day 57 and 141
  Forced expiratory volume in 1 second (FEV1) is the volume exhaled during the first second of a forced expiratory maneuver started from the level of total lung capacity. Spirometry testing must be performed in the morning between 6 11 am according to the schedule of study procedures. After the first screening spirometry completed, the
Proportion of the number of AE reporting (incidence of adverse event) | 12 weeks follow up
  AE

OTHER OUTCOMES:
Change in IL-6 | during the study (8 weeks treatment period and 12 weeks follow up
  IL-6

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Ho, Director, Study Director — Oneness Biotech
Locations (9):
- Taiwan (9):
  - NTUH Hsin-Chu Branch, Hsinchu
  - Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City
  - China Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Taiwan University Hospital, Taipei
  - Taipei Medical University Hospital, Taipei
  - Taipei Medical University-Shuang Ho Hospital,Ministry of Health and Welfare, Taipei
  - Taipei Municipal Wanfang Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei